CLINICAL TRIAL: NCT02072538
Title: Role of Pre-discharge vs. Early Post-discharge Stress Testing and Implementation of the GRACE Risk Score for Safe Discharge of Patients With an ACS and a Negative High Sensitivity Troponin T Result Within 3 Hours After Presentation to a Chest Pain Unit
Brief Title: Pre-discharge vs. Early Post-discharge Stress Testing and GRACE Score for Safe Discharge of ACS-patients With a Negative Hs-troponin T Result
Status: Withdrawn | Type: Observational
Why Stopped: no Sponsor
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Professor Hugo Katus, Head of Cardiology, University Hospital Heidelberg
Other Study IDs: UHHD-BM-002
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Major Adverse Cardiovascular Events; Troponin T; GRACE Score
Keywords: Stress testing; Troponin T; GRACE score; Outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre-discharge stress testing: Stress-testing (e.g. treadmill exercise test, stress-echochardiography)
- Post-discharge stress testing: Stress-testing (e.g. treadmill exercise test, stress-echochardiography)

SUMMARY:
New high-sensitivity cardiac troponin (hs-cTn) assays allow earlier detection of acute myocardial infarction (AMI). Furthermore, elevated values were associated with an increased risk of recurrent AMI or death. Therefore, guidelines recommend an early invasive strategy in patients with elevated admission values and kinetic changes. Other criteria for an early invasive strategy include a GRACE risk score >140 points or other cardiovascular risk factors. Hs-cTn assays allow discrimination of patients at very low and high risk. Studies confirmed safety of early discharge protocols in patients with unstable angina (UAP). The aim of this study is to 1) confirm the safety of early discharge without invasive strategy in patients with UAP and to 2) review the optimal timing of stress-testing. Therefore, patients are being randomized into 2 groups with pre-discharge and early post-discharge stress-testing. Endpoints are major adverse cardiovascular events within 30 and 90 days.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting to the emergency department ("chest pain unit")
* typical angina pectoris
* absence of symptoms since presentation
* at least 18 years
* low GRACE risk score (<140 points)
* informed consent, signed agreement

Exclusion Criteria:

* conditions with need for immediate workup
* mental disorders
* dementia
* pregnancy, breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to our emergency department ("chest pain unit") with typical angina pectoris are being screened for participation. Those meeting the inclusion criteria (typical angina pectoris, absence of symptoms since presentation, low GRACE risk score) are included.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular event | 30 days

SECONDARY OUTCOMES:
Major adverse cardiovascular event | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Giannitsis, MD, Principal Investigator — University Hospital Heidelberg; Hugo A Katus, MD, Study Chair — University Hospital Heidelberg
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany